CLINICAL TRIAL: NCT05882123
Title: Gender Heterogeneity in the Influencing Factors for Cerebral Microbleeds in Acute Ischemic Stroke Patients
Status: Completed | Type: Observational
Sponsor: Xin Guo (Other)
Responsible Party: Sponsor-Investigator, Xin Guo, Attending physician, The First Hospital of Hebei Medical University
Organization: The First Hospital of Hebei Medical University (Other)
Other Study IDs: 20220642
Record Dates: First submitted 2023-05-11; First posted 2023-05-31 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Acute Ischemic Stroke
Keywords: Acute ischemic stroke; Cerebral microbleeds; Influencing factors; Gender heterogeneity
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Comparison of clinical data between AIS patients in CMB and non-CMB groups
- without CMBs; with CMBs
  Interventions: Other: cerebral microbleeds
- male; female
  Interventions: Other: cerebral microbleeds

INTERVENTIONS:
Other: cerebral microbleeds — Whether patients with acute ischemic stroke are complicated by cerebral microbleeds
  Groups: male; female; without CMBs; with CMBs

SUMMARY:
The investigators continuously collected data from 482 AIS inpatients at the Neurology Department of Hebei General Hospital. Both demographic and clinical data were collected from the study subjects. Different head magnetic resonance imaging sequences were used to assess the subjects' CMBs, white matter lesions, and old lacunar infarcts (LI). Various statistical methods, including the t-test, χ2 test, and logistic regression, were used to analyze the gender heterogeneity of the influencing factors for CMBs in AIS patients.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years and older
* Must meet the diagnostic criteria for AIS as presented in the Chinese Guidelines for Diagnosis and Treatment of Acute Ischemic Stroke 2014
* Must be in good physical condition and have the ability to cooperate with MRI examinations
* Must have underwent SWI

Exclusion Criteria:

* MRI contraindications present, such as cardiac pacemaker, cardiac stents, or metal implants
* Head MRI or carotid artery ultrasound suggests the presence of severe stenosis or occlusion in the intracranial or extracranial segments of the cerebral arteries
* Severe comorbid diseases, such as cardiac, pulmonary, hepatic, and renal insufficiencies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In this study, the data of patients with AIS who were admitted to the Department of Neurology of Hebei Provincial People's Hospital from January 2014 to December 2015 were continuously collected.
Sampling Method: Non-Probability Sample
Enrollment: 482 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Comparison of clinical data between AIS patients in CMB and non-CMB groups | from January 2014 to December 2015
  Differences in general information between AIS patients in CMB and non-CMB groups
Comparison of clinical data between male and female AIS patients | from January 2014 to December 2015
  Differences in general informationbetween male and female AIS patients
Comparison of CMB-related characteristics between the male and female AIS patients | from January 2014 to December 2015
  Differences in CMB-related characteristics between the male and female AIS patients
Predictive factor analysis for CMBs in male AIS patients | from January 2014 to December 2015
  CMB-related factors in male AIS patients
Predictive factor analysis for CMBs in female AIS patients | from January 2014 to December 2015
  CMB-related factors in female AIS patients

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Guo X, Xing Y, Teng Z, Shen Z, Guo X, Lv P, Tian S. Gender heterogeneity in the influencing factors for cerebral microbleeds in acute ischemic stroke patients. Curr Med Res Opin. 2023 Jul;39(7):1045-1054. doi: 10.1080/03007995.2023.2219581. Epub 2023 Jun 20. PMID 37259500